CLINICAL TRIAL: NCT05152576
Title: A Phase 2, Multicenter, Randomized, Placebo-controlled Study to Evaluate the Safety and Efficacy of OnabotulinumtoxinA X for Forehead Lines
Brief Title: A Study To Assess the Adverse Effects and Change in Condition of OnabotulinumtoxinA X Injection in Adult Participants With Forehead Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M21-606
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Forehead Lines
Keywords: Forehead Lines; OnabotulinumtoxinA X

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo will be injected into the forehead on Day 1.
  Interventions: Drug: Placebo
- OnabotulinumtoxinA X Dose A (Experimental): OnabotulinumtoxinA X will be injected into the forehead on Day 1.
  Interventions: Drug: OnabotulinumtoxinA X
- OnabotulinumtoxinA X Dose B (Experimental): OnabotulinumtoxinA X will be injected into the forehead on Day 1.
  Interventions: Drug: OnabotulinumtoxinA X
- OnabotulinumtoxinA X Dose C (Experimental): OnabotulinumtoxinA X will be injected into the forehead on Day 1.
  Interventions: Drug: OnabotulinumtoxinA X

INTERVENTIONS:
Drug: OnabotulinumtoxinA X — Intramuscular Injection
  Other Names: OnabotA X
  Arms: OnabotulinumtoxinA X Dose A; OnabotulinumtoxinA X Dose B; OnabotulinumtoxinA X Dose C
Drug: Placebo — Intramuscular Injection
  Arms: Placebo

SUMMARY:
Facial lines that develop from repeated facial expression, such as forehead lines (FHL), are typically treated by selectively weakening specific muscles with small quantities of botulinum toxin. OnabotulinumtoxinA X is being investigated as another form of treatment to treat FHL by inhibiting the release of the neurotransmitter that causes the overactivity of the muscles responsible for the severity of these facial lines. The purpose of this study is to evaluate the safety and change in condition of 3 doses of OnabotulinumtoxinA X for the treatment of moderate to severe forehead lines.

Study doctors will determine if a subject is eligible for the study. If so, the subject will be randomized into 1 of the 4 groups, called treatment arms. There is a 1 in 4 chance that a participant will be assigned to placebo. Around 120 adult participants with FHL will be enrolled in the study in approximately 10 sites in the United States.

Participants will receive either intramuscular injections of onabotulinumtoxinA X or placebo.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular monthly visits during the study at the study site.

ELIGIBILITY:
Inclusion Criteria:

* Participant has sufficient visual acuity without the use of eyeglasses (contact lens use is acceptable) to accurately assess their facial lines
* Participant has moderate or severe Forehead Lines (FHL) at maximum eyebrow elevation

Exclusion Criteria:

* History of known immunization to any botulinum toxin serotype.
* History of known hypersensitivity to any botulinum toxin serotype, or any other constituents of the study drug or its excipients, and/or other products in the same class.
* Presence or history of any medical condition that may place the participant at increased risk following exposure to OnabotulinumtoxinA X or interfere with the study evaluation, including:

Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function.

* History of Facial nerve palsy.
* Infection or dermatological condition at the site of study drug injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (8):
- United States (8):
  - The Eye Research Foundation /ID# 241512, Newport Beach, California
  - Steve Yoelin MD Medical Associate Inc /ID# 239771, Newport Beach, California
  - The Center for Dermatology Cosmetics & Laser Surgery /ID# 239776, Mount Kisco, New York
  - Skin Search of Rochester Inc. /ID# 239773, Rochester, New York
  - Dermatology Consulting Service /ID# 239779, High Point, North Carolina
  - Wilmington Dermatology Center /ID# 239778, Wilmington, North Carolina
  - Dallas Plastic Surgery Institute /ID# 239777, Dallas, Texas
  - Duplicate_Austin Institute for Clinical Research /ID# 239783, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
Started | 30 | 35 | 31 | 28
Completed | 25 | 34 | 31 | 26
Not Completed | 5 | 1 | 0 | 2
Not completed — Lost to Follow-up | 3 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Other | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C | Total
Number analyzed (Participants) | 30 | 35 | 31 | 28 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (12.33) | 43.7 (11.97) | 46.6 (11.82) | 50.5 (12.87) | 46.6 (12.32)
Age, Customized [Count of Participants; unit: Participants]
  18-25 | 1 | 2 | 2 | 0 | 5
  26-40 | 9 | 11 | 7 | 8 | 35
  41-55 | 11 | 16 | 13 | 9 | 49
  56-64 | 8 | 5 | 9 | 7 | 29
  >=65 | 1 | 1 | 0 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 28 | 26 | 108
  Male | 4 | 7 | 3 | 2 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 4 | 6 | 19
  Not Hispanic or Latino | 24 | 32 | 27 | 22 | 105
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 30 | 34 | 28 | 26 | 118
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a casual relationship with this treatment. The investigator assesses the relationship of each event to the use of the study. A serious adverse event (SAE) is an event that results in death, is life threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event, that based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Time Frame: Day 1 to Day 180
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
Number analyzed (Participants) | 29 | 35 | 31 | 28
Participants | 10 | 12 | 18 | 13

2. Primary Outcome: Percentage of Participants With Potentially Clinically Significant Vital Sign Parameters
Description: Percentage of participants with potentially clinically significant vital sign measurements like systolic and diastolic blood pressure will be assessed.
Time Frame: Day 1 to Day 180
Population: Safety population
  Overall Number of Participants Analyzed = Except for Temperature, number of subjects with an available baseline value and at least 1 postbaseline assessment; for Temperature, number of subjects with at least 1 postbaseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
Number analyzed (Participants) | 29 | 35 | 31 | 27
Participants
  Systolic Blood Pressure (mmHg): ≥ 160 and Increase of ≥ 20 | 0 | 1 | 1 | 1
  Systolic Blood Pressure (mmHg): ≤ 90 and Decrease of ≥ 20 | 0 | 1 | 1 | 0
  Diastolic Blood Pressure (mmHg): ≥ 100 and Increase of ≥ 15 | 1 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg): ≤ 50 and Decrease of ≥ 15 | 0 | 0 | 0 | 0
  Heart Rate (beats/min): ≥ 110 and Increase of ≥ 15 | 0 | 0 | 0 | 0
  Heart Rate (beats/min): ≤ 50 and Decrease of ≥ 15 | 0 | 0 | 0 | 0
  Temperature (C): ≥ 38.3 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Achievement of ≥ 1-grade Improvement From Baseline on the Investigator-rated Clinician Forehead Lines Scale at Maximum Contraction.
Description: Facial Wrinkle Scale - Forehead Lines (FWS-FHL) at maximum contraction (also known as eyebrow elevation)
  The Clinician Forehead Lines Scale is a four point scale used to assess the severity of forehead lines at maximum contraction ranging from 0 - None to 3 - Severe.
Time Frame: Day 1 to Day 30
Population: Intent-to-Treat Population
  Overall Number of Participants Analyzed = Number of subjects with data at baseline and the visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
Number analyzed (Participants) | 29 | 34 | 31 | 27
percentage of participants | 58.6 [40.7 to 76.5] | 100 [100 to 100] | 96.8 [90.6 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Placebo vs OnabotulinumtoxinA X Dose A; Confidence interval for responder rate is calculated using normal approximation; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline investigator-rated FWS-FHL at maximum; Rate Difference = 41.4, 95% CI 2-sided [23.5 to 59.3]
Statistical Analysis 2: Comparison: Placebo vs OnabotulinumtoxinA X Dose B; Confidence interval for responder rate is calculated using normal approximation; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline investigator-rated FWS-FHL at maximum; Rate Difference = 38.2, 95% CI 2-sided [19.2 to 57.1]
Statistical Analysis 3: Comparison: Placebo vs OnabotulinumtoxinA X Dose C; Confidence interval for responder rate is calculated using normal approximation; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline investigator-rated FWS-FHL at maximum; Rate Difference = 41.4, 95% CI 2-sided [23.5 to 59.3]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the end of the study. The median time on follow-up was 190, 190, 191, and 189 days for Placebo, OnabotulinumtoxinA X Dose A, Dose B and Dose C, respectively.
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/35 | 0/31 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/35 | 0/31 | 0/28
Other Adverse Events (participants affected / at risk) | 4/30 | 5/35 | 10/31 | 9/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | OnabotulinumtoxinA X Dose A (N=35) | OnabotulinumtoxinA X Dose B (N=31) | OnabotulinumtoxinA X Dose C (N=28)
KIDNEY INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | OnabotulinumtoxinA X Dose A (N=35) | OnabotulinumtoxinA X Dose B (N=31) | OnabotulinumtoxinA X Dose C (N=28)
EYELID PTOSIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
INJECTION SITE BRUISING (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
INJECTION SITE PAIN (General disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
INJECTION SITE SWELLING (General disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
ASYMPTOMATIC COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 4 (4) | 5 (5) | 3 (3)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT05152576/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT05152576/SAP_001.pdf